CLINICAL TRIAL: NCT02856711
Title: Assessing the CenteringPregnancy Planning to Parent Innovation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: Doris Duke Charitable Foundation (Other)
Responsible Party: Principal Investigator, Morgan Brockington, Health Outreach & Evaluation Coordinator, Vital Village Network, General Pediatrics, Boston Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: H-34199
Record Dates: First submitted 2016-04-25; First posted 2016-08-05 (Estimated); Last update posted 2016-11-23 (Estimated); Status verified 2016-11

CONDITIONS: Stress, Psychologic; Pregnancy
Keywords: Group Prenatal Visits,CenteringPregnancy
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Trauma-informed group (Experimental): These groups will use the enhanced Centering Pregnancy curriculum.
  Interventions: Behavioral: Trauma-informed group
- Control group (No Intervention): These groups will use the standard CenteringPregnancy curriculum.

INTERVENTIONS:
Behavioral: Trauma-informed group — The two interventions will be: 1) A viewing of "All Babies Cry" and a discussion of what it's like to be a new parent, 2) A "Planning to Parent" stress activity where parents discuss when they have felt overwhelmed, the coping mechanisms they used, and what can be done to manage those emotions in the future. The goal of this project is to gain insight from current participants in CenteringPregnancy group care around the ways that these interventions can better prepare parents to deal with the common stresses of parenthood.
  Arms: Trauma-informed group

SUMMARY:
The investigators propose to evaluate how the CenteringPregnancy curriculum compared with an enhanced curriculum, with the addition of 2 trauma-informed interventions, affects how new parents prepare for parenting and respond to common stressors.

DETAILED DESCRIPTION:
The two interventions will be 1) A viewing of "All Babies Cry" and a discussion of what it's like to be a new parent and 2) A "Planning to Parent" stress activity where parents discuss when they have felt overwhelmed, the coping mechanisms they used, and what can be done to manage those emotions in the future. The goal of this project is to gain insight from current participants in CenteringPregnancy group care around the ways that these interventions can better prepare parents to deal with the common stresses of parenthood.

The investigators will assess the curriculum by administering pre-test and post-test surveys to CenteringPregancy patients within 6 groups. Three of the groups will use the regular CenteringPregnancy curriculum and 3 of the groups will use the enhanced Centering Pregnancy curriculum. Participants will be recruited to CenteringPregnancy, and thus this study, as part of Boston Medical Center Obstetrics/Gynecology Associate's regular prenatal registration process and will be assigned to prenatal groups based on due date. The informed consent and pre-test will be administered to patients at Session 7 of the CenteringPregnancy curriculum and the post-test will be administered to patients at the postpartum visit. The control CenteringPregnancy groups will follow the regular curriculum as written in the CenteringPregnancy Facilitator's Guide. The experimental CenteringPregnancy groups will follow the regular CenteringPregnancy curriculum, with the addition of the "All Babies Cry" intervention during Session 7 (30-34 weeks) and the "Planning to Parent" stress intervention during Session 8 (32-36 weeks). There will be no individual interviews of participants. Following the postpartum survey, the Research Assistant will conduct electronic medical record chart reviews of the study participants.

The investigators propose to seek between 24 and 36 patients for the 3 control groups and between 24 and 36 patients for the 3 experimental groups, for a total of 48-72 subjects. Pre-test and post-test surveys will be collected by a member of the research team. Surveys will be kept in a locked desk and will later analyzed. The intent of this study is to gather important information on ways to improve group-based prenatal care from a patient-centered, trauma-informed perspective. This will ultimately help to improve both family and child well being and reduce the risk of child abuse, neglect and parental and toxic stress in the greater Boston area.

ELIGIBILITY:
Inclusion Criteria:

* Fluent in English language. Able to complete a written survey in English.
* Currently participating in CenteringPregnancy groups at Boston Medical Center.
* A woman at least 18 years old or older.

Exclusion Criteria:

* Women who do not attend the sessions where the intervention are conducted
* Women <18 years old will not be recruited. All participants will be 18 years old or older.
* Not fluent in English language.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2015-11; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Sources of parenting information | 1 month postpartum
Types of parenting support used | 1 month postpartum
Types of parental behaviors demonstrated | 1 month postpartum
Frequency of depressed moods (scale) | 1 month postpartum
Parents' levels of social support | 1 month postpartum
Frequency of parenting stress (scale) | 1 month postpartum

OTHER OUTCOMES:
Gestational age at first prenatal visit | 1 month postpartum
Number of prenatal visits | 1 month postpartum
Gestational age at delivery | 1 month postpartum
Birth weight | 1 month postpartum
Delivery Mode | 1 month postpartum
Neonatal intensive care unit admission | 1 month postpartum
Breastfeeding rate (scale) | 1 month postpartum
Body mass index | 1 month postpartum
Contraceptive plan | 1 month postpartum
Contraceptive method used | 1 month postpartum
Sexually transmitted disease exposure | 1 month postpartum
Tobacco use | 1 month postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Beth Monahan, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided